CLINICAL TRIAL: NCT04170790
Title: Evaluation of Drug Interactions of Saxagliptin With Sildenafil in Healthy Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Yousri Mansour, Masters Of Clinical Pharmacy- faculty of Pharmacy- Ain shams University, Ain Shams University
Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 57
Record Dates: First submitted 2019-11-14; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus, Type 2; Erectile Dysfunction With Diabetes Mellitus; Drug Interaction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Eighteen healthy volunteers will be recruited in Sequential, single center study to determine pharmacokinetic parameters of Saxagliptin, and sildenafil,(AUC0→∞), (AUC0→t); Cmax; tmax; t½, k; ka) will be measured using validated LC-MS/MS method. Therapeutic doses will be given to volunteers as follows: Sildenafil 50 mg single dose on day 1, then washout period from day 2 till day 8. Saxagliptin 5 mg once/day will be given from day 9 till day 12, then on day 13 the two drugs will be co-administered. Blood samples (5ml) for pharmacokinetic analysis will be collected on days 1 and 13 for Sildenafil as well as on days 12 and 13 for Saxagliptin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteer (Experimental): Day 1: Sildenafil 50 mg single dose Day 2-Day 8: Washout period Day 9-12: Saxagliptin 5 mg Once/day Day 13: Sildenafil 50 mg+ Saxagliptin 5 mg
  Interventions: Drug: Saxagliptin 5mg; Drug: Sildenafil 50 mg

INTERVENTIONS:
Drug: Saxagliptin 5mg — Saxagliptin 5mg oral tablet
  Other Names: Onglyza
Drug: Sildenafil 50 mg — Sildenafil 50 mg Oral Tablet
  Other Names: Viagra

SUMMARY:
Patients with diabetes are three times more likely to develop erectile dysfunction (ED), and longer duration of diabetes is strongly associated with ED. The possibility of pharmacokinetic interactions may occur as the two drugs are metabolized by hepatic CYP3A4 and their co administration may affect their plasma concentrations. the aim of work is to investigate the effect of sildenafil a CYP3A4 substrate and inhibitor on the pharmacokinetics and safety of Saxagliptin, a CYP3A4 substrate Subjects and Methods: Eighteen healthy volunteers will be recruited in Sequential, single center study to determine pharmacokinetic parameters of Saxagliptin, and sildenafil,(AUC0→∞), (AUC0→t); Cmax; tmax; t½, k; ka) will be measured using validated LC-MS/MS method. Therapeutic doses will be given to volunteers as follows: Sildenafil 50 mg single dose on day 1, then washout period from day 2 till day 8. Saxagliptin 5 mg once/day will be given from day 9 till day 12, then on day 13 the two drugs will be co-administered. Blood samples (5ml) for pharmacokinetic analysis will be collected on days 1 and 13 for Sildenafil as well as on days 12 and 13 for Saxagliptin.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years.
2. Ideal weight within the normal range according to accepted life tables.
3. Non-contributory history and normal physiological examination.
4. Laboratory data within normal limits.
5. Performance and compliance.
6. The subjects should be without known history of alcohol or drug abuse problems and should preferably be non-smokers.
7. The volunteers will be asked to provide a complete medical history, and complete a physical examination, laboratory tests (hematology, clinical chemistry, urinalysis serology (including hepatitis B surface antigen, anti-hepatitis C virus and antihuman immunodeficiency virus antibody).

Exclusion Criteria:

1. A known hypersensitivity to the drug.
2. Gastrointestinal diseases.
3. Auto immune diseases.
4. Renal diseases or dysfunction.
5. Cardiovascular disease of any type.
6. Pancreatic disease including diabetes.
7. Hepatic disease.
8. Hematological, osteopathic, or pulmonary disease.
9. History of alcoholism or drug abuse.
10. Serious Psychological illness.
11. Positive HIV-I.
12. Smoking (if including they should be identified).
13. Abnormal (out of range) laboratory values.
14. Subject who have taken any medication (Rx or OTC) less than two weeks of the trials starting date.
15. Subject who have donated blood or who have been in multiple dosing studies requiring a large volume of blood (more than 500 ml) to be drawn within six weeks preceding the start of the trials.
16. Any prior surgery of the gastrointestinal tract that may interfere with drug absorption.
17. Treatment with any known enzyme-inducing / inhibiting agents within 30 days prior to the start of the study and throughout the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 18, and 24 hours post-dose.
  Maximum Plasma Concentration
(AUC0→∞) | pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 18, and 24 hours post-dose.
  Area Under Curve Infinity
(AUC0→t) | pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 18, and 24 hours post-dose.
  Area Under the Curve
tmax; | pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 18, and 24 hours post-dose.
  Time to reach Maximum concentration
T½ | pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 18, and 24 hours post-dose.
  Drug half Life
Ke | pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 18, and 24 hours post-dose.
  Elimination Rate
ka | pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 18, and 24 hours post-dose.
  Absorption Rate
Blood Pressure | measured before dosing and at 2, 4, 6, 8, and 10 hours after drug administration on each day of blood sampling
  changes in Systolic and Diastolic Blood Pressure from normal range
Heart Rate | measured before dosing and at 2, 4, 6, 8, and 10 hours after drug administration on each day of blood sampling
  Changes in heart rate from normal range

REFERENCES:
- [Derived] Mansour RY, ElBorolossy R, Shaheen SM, Sabri NA. Evaluation of drug interactions of saxagliptin with sildenafil in healthy volunteers. Eur J Clin Pharmacol. 2022 Dec;78(12):1935-1944. doi: 10.1007/s00228-022-03397-w. Epub 2022 Oct 10. PMID 36214883